CLINICAL TRIAL: NCT00050427
Title: A Phase 2 Study of ET-743 in Subjects With Advanced Breast Cancer
Brief Title: A Study of ET-743 (Trabectedin) in Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sr Dir Clinical Research, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004525; ET743-INT-3; NCT01328327 (obsolete NCT alias)
Record Dates: First submitted 2002-12-09; First posted 2002-12-18 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Breast Neoplasms; Neoplasms; Neoplasms by Site; Breast Diseases; Skin Diseases
Keywords: Trabectedin; Yondelis; ET743; Advanced breast cancer; Breast; Cancer; Antineoplastic Agents, Alkylating Agents; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasms by Site; Breast Diseases; Skin Diseases | interventions — Trabectedin

ARMS (2):
- 001 (Experimental): ET743 580 mcg/m2 3-hour i.v. infusion on Days 1 8 and 15 every 28 days for up to approximately 52 weeks in the absence of disease progression. Dexamethasone 10 mg i.v will be administered 30 minutes prior to each trabectedin infusion.
  Interventions: Drug: ET743
- 002 (Experimental): ET743 1 300 mcg/m2 3 hour i.v. infusion once every 21 days for up to approximately 52 weeks in the absence of disease progression. Dexamethasone 10 mg i.v will be administered 30 minutes prior to each trabectedin infusion.
  Interventions: Drug: ET743

INTERVENTIONS:
Drug: ET743 — 580 mcg/m2, 3-hour i.v. infusion, on Days 1, 8, and 15 every 28 days for up to approximately 52 weeks in the absence of disease progression. Dexamethasone, 10 mg i.v, will be administered 30 minutes prior to each trabectedin infusion.
  Arms: 001
Drug: ET743 — 1,300 mcg/m2, 3 hour i.v. infusion once every 21 days for up to approximately 52 weeks in the absence of disease progression. Dexamethasone, 10 mg i.v, will be administered 30 minutes prior to each trabectedin infusion.
  Arms: 002

SUMMARY:
The purpose of this study is to test the safety and effectiveness of an investigational chemotherapy agent in patients with advanced breast cancer.

DETAILED DESCRIPTION:
Patients will be enrolled in the study after all study specific-entry criteria are met and informed consent is obtained. Patients will be required to attend regular clinic visits to receive study medication and have their status monitored. Patients will also be required to have radiologic tumor assessments performed at multiple times throughout the study. A detailed explanation can be provided by the study physician (Investigator) conducting this study. Trabectedin 580 mcg/m2 once weekly for 3 consecutive weeks (Treatment A) or 1,300 mcg/m2 once every 21 days (Treatment B) will be given to patients as a 3-hour intravenous (i.v). infusion via a central venous catheter which is a tube placed into a large vein that is used to administer medications. All patients will be given dexamethasone 10 mg i.v. 30 minutes before each trabectedin infusion. Patients may receive multiple cycles of trabectedin in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced breast cancer
* Prior therapy with anthracycline and taxane (2 types of chemotherapy drugs)
* At least one measureable tumor lesion
* Adequate bone marrow, hepatic and renal function
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1

Exclusion Criteria:

* Known hypersensitivity to any components of the i.v. formulation of ET-743 or dexamethasone
* Pregnant or lactating women
* Known metastases (spread) of cancer to the central nervous system
* History of another neoplastic disease unless in remission for five years or more.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2002-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with objective response in each treatment arm. | Up to approximately 52 weeks

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 52 weeks
Time to progression (TTP) | Up to approximately 52 weeks
Overall survival (OS) | Up to approximately 52 weeks
The number of patients with treatment-emergent adverse events | Up to approximately 52 weeks
Concentrations of trabectedin in plasma as a measure of the pharmacokinetics of trabectedin | During the first two 28-day treatment cycles

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Goldstein LJ, Gurtler J, Del Prete SA, Tjulandin S, Semiglazov VF, Bayever E, Michiels B. Trabectedin as a single-agent treatment of advanced breast cancer after anthracycline and taxane treatment: a multicenter, randomized, phase II study comparing 2 administration regimens. Clin Breast Cancer. 2014 Dec;14(6):396-404. doi: 10.1016/j.clbc.2014.06.006. Epub 2014 Aug 15. PMID 25239225